CLINICAL TRIAL: NCT03179280
Title: Effect of Dual-wave Insulin Bolus on Postprandial Glycaemia According to the Composition of the Meal in Adolescents With Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion
Brief Title: Effect of Dual-wave Insulin Bolus on Postprandial Glycaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Assimina Galli-Tsinopoulou, Associate Professor, 4th Department of Pediatrics, Medical School of Aristotle University of Thessaloniki, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Dual-wave insulin
Record Dates: First submitted 2017-05-04; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Type1 Diabetes
Keywords: Type 1 diabetes; Dual-wave bolus; Postprandial euglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adolescents with T1D on CSII (Active Comparator): 3 standard meals with varying composition were consumed and combined with alternative types of D/WB and S/WB All participants used the rapid-acting insulin analogue aspart (NovoRapid®, Novonordisk A/S, Bagsvaerd, Denmark) and total insulin dose administered to each one for each test meal was known in advance, according to the insulin to carbohydrate ratio that had been calculated during the 2-week pre-study period.
  Interventions: Drug: insulin
- Healthy adolescents (No Intervention): 3 standard meals with varying composition were consumed

INTERVENTIONS:
Drug: insulin — All participants used the rapid-acting insulin analogue aspart (NovoRapid®, Novonordisk A/S, Bagsvaerd, Denmark) and total insulin dose administered to each one for each test meal was known in advance, according to the insulin to carbohydrate ratio that had been calculated during the 2-week pre-study period.
  Other Names: NovoRapid
  Arms: Adolescents with T1D on CSII

SUMMARY:
A study was conducted in adolescents with type 1 diabetes (T1D) examining the effect of different bolus types on 6-h postprandial glucose levels after the consumption of 3 standard meals with varying composition. Participants were asked to consume 10 different combinations of meal and bolus type.

DETAILED DESCRIPTION:
The nutritional recommendations of children and adolescents with T1D should be similar to those of healthy people in order to achieve the desirable growth. Not only the carbohydrates' intake is underlined according to special guidelines by Canadian diabetes association, American diabetes association and International Society for Paediatric and Adolescent Diabetes but also proteins and fats are suggested to be taken into consideration in the management of T1D. In order to reach the desirable euglycemic control, children and adolescents can use multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII). By using the CSII the insulin can be administrated in three different patterns; as a normal bolus, as a dual wave bolus and as a square wave bolus. Dual wave insulin bolus (D/WB) is suggested as the most suitable option based on the effects that is having after meals with different content of carbohydrates, fats and proteins. The aim of this study was to evaluate the impact of different types of D/WB on PPG after 3 given meals, in adolescents with T1D on CSII. In order to achieve that, 3 different meals were designed and combined with alternative types of boluses, D/WB and square wave insulin bolus (S/WB).

ELIGIBILITY:
Inclusion Criteria:

* duration of T1D >3 years, CSII therapy for at least 1 year, good to moderate glycaemic control, as evidenced by HbA1c levels <8.5% (69 mmol/mol).

Exclusion Criteria:

* Subjects with eating disorders, food allergy, celiac disease and known diabetic complications

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
post-prandial euglycaemia (PPG) | 3 days
  the impact of different types of D/WB on PPG after three given meals, in adolescents with T1D on CSII. In order to achieve that, three different meals were designed and combined with alternative types of boluses, D/WB and S/WB

CONTACTS AND LOCATIONS:
Overall Officials: Assimina Galli-Tsinopoulou, Ass Prof, Study Chair — Unit of Pediatric Endocrinology, Diabetes and Metabolism-4th Department of Pediatrics, Medical School of Aristotle University of Thessaloniki
Locations (1):
- Unit of Pediatric Endocrinology, Diabetes and Metabolism-4th Department of Pediatrics, Medical School of Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heinemann L. Insulin pump therapy: what is the evidence for using different types of boluses for coverage of prandial insulin requirements? J Diabetes Sci Technol. 2009 Nov 1;3(6):1490-500. doi: 10.1177/193229680900300631. PMID 20144405
- [Result] Chase HP, Saib SZ, MacKenzie T, Hansen MM, Garg SK. Post-prandial glucose excursions following four methods of bolus insulin administration in subjects with type 1 diabetes. Diabet Med. 2002 Apr;19(4):317-21. doi: 10.1046/j.1464-5491.2002.00685.x. PMID 11943004
- [Result] Lee SW, Cao M, Sajid S, Hayes M, Choi L, Rother C, de Leon R. The dual-wave bolus feature in continuous subcutaneous insulin infusion pumps controls prolonged post-prandial hyperglycaemia better than standard bolus in Type 1 diabetes. Diabetes Nutr Metab. 2004 Aug;17(4):211-6. PMID 15575341